CLINICAL TRIAL: NCT00785200
Title: MRSA Colonization and Control in the Dallas County Jail
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: University of Texas Southwestern Medical Center (Other); Sage Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14633A (R01 CI000373-03); R01CI000373-03 (NIH)
Record Dates: First submitted 2008-11-03; First posted 2008-11-05 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2010-02

CONDITIONS: Methicillin-resistant Staphylococcus Aureus; Skin Diseases, Infectious; Soft Tissue Infections
Keywords: MRSA; Methicillin-resistant Staphylococcus aureus; Chlorhexidine; Asymptomatic colonization; Asymptomatic colonization, MRSA; Skin and soft tissue infections
MeSH Terms: conditions — Skin Diseases, Infectious; Soft Tissue Infections; Asymptomatic Infections | interventions — Chlorhexidine; Water

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Chlorhexidine (Experimental): Approximately 500 detainees housed in approximately 23 detention tanks will be enrolled and receive 2% chlorhexidine-soaked disposable wash cloths (Sage Products, Inc.) to clean their skin on Mondays, Wednesdays, and Fridays for 6 months. Newly arrived detainees in the tanks will be offered enrollment in the study on a biweekly schedule.
  Interventions: Other: Chlorhexidine
- Water (Placebo Comparator): Approximately 500 detainees in approximately 23 detention tanks will receive water-soaked wash cloths to clean their skin each Monday, Wednesday, and Friday for a 6-month period. If detainees newly arrive to these study tanks, they will be offered enrollment on a biweekly schedule.
  Interventions: Other: Water
- Usual care (No Intervention): Approximately 500 detainees in approximately 23 detention tanks will be enrolled. These detainees will not receive any intervention. They will be followed for 6 months, and newly arrived detainees will be offered enrollment on a biweekly schedule.

INTERVENTIONS:
Other: Chlorhexidine — Chlorhexidine-soaked disposable cloths will be distributed each Monday, Wednesday, and Friday to each enrolled detainee for a 6-month period.
  Arms: Chlorhexidine
Other: Water — Water-soaked disposable wash cloths identical in appearance to the CHG cloths will be distributed to enrolled detainees on every Monday, Wednesday, and Friday for a 6-month period.
  Arms: Water

SUMMARY:
The goal of this 3-year project is to control the spread of community-associated methicillin-resistant Staphylococcus aureus (CA-MRSA) in the Dallas County Jail. CA-MRSA is a bacterium spreading rapidly through healthy populations and becoming an epidemic in many regions of the U.S. Many people in the community are asymptomatically colonized by MRSA. There have been outbreaks of MRSA infections at prisons and jails. We will study the spread of MRSA in the jail to better understand how the bacteria are transmitted from person to person there and how we can prevent their transmission. All detainees asked to participate must give informed consent to do so; their privacy will be carefully protected. Detainees with a history of allergy to CHG will be excluded. Seventeen objects in the jail will be sampled for contamination with MRSA. Bacteria will be collected from all cultures obtained from patients with bacterial skin infections for 18 months in a part of the jail in order to determine how frequently these infections are caused by MRSA relative to other bacteria. A group of about 1500 adult detainees will be tested for colonization with MRSA in order to determine how commonly detainees carry the bacterium. A cluster-randomized 6-month study will be undertaken among these detainees and those who take their places when they leave the jail to determine if chlorhexidine (CHG)-containing disposable wash cloths for skin cleaning can decrease the prevalence of MRSA skin or nose colonization. Detainees receiving CHG cloths (about 500 detainees) will be compared to detainees receiving water-soaked cloths for skin cleaning (about 500 detainees) or no intervention (about 500 detainees). The primary outcome will be a difference in average colonization prevalence in detention tanks, which are discrete detention units housing detainees, comparing the usual care to the CHG-exposed tanks after 6 months of CHG cloth use. A secondary outcome will be a decrease in skin infections from any cause in the tanks receiving CHG compared with usual care. All of the MRSA isolates and a sample of the S. aureus isolates susceptible to methicillin from specimens colonizing or infecting detainees, as well as those contaminating surfaces and objects in the jail will be tested genetically in order to determine which strains of MRSA are present in the jail. This study may identify ways to stop the spread of MRSA among people in jails and prisons, as well as other places.

ELIGIBILITY:
Inclusion Criteria:

* Admission to a participating tank in the jail

Exclusion Criteria:

* History of hypersensitivity reaction to chlorhexidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4194 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Average prevalence of MRSA hand or nasal colonization in study tanks (i.e., 24-60-person detention divisions) receiving CHG cloths vs. usual care | 6 months

SECONDARY OUTCOMES:
Average incidence of skin and soft tissue infections requiring incision and drainage per tank in a 6 month period, comparing group of study tanks receiving CHG-soaked washcloths to those receiving usual care. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Daum, MD, Principal Investigator — University of Chicago
Locations (1):
- The Dallas County Jail, Dallas, Texas, United States

REFERENCES:
- [Derived] David MZ, Siegel JD, Henderson J, Leos G, Lo K, Iwuora J, Porsa E, Schumm LP, Boyle-Vavra S, Daum RS. A randomized, controlled trial of chlorhexidine-soaked cloths to reduce methicillin-resistant and methicillin-susceptible Staphylococcus aureus carriage prevalence in an urban jail. Infect Control Hosp Epidemiol. 2014 Dec;35(12):1466-73. doi: 10.1086/678606. PMID 25419768